CLINICAL TRIAL: NCT01728545
Title: The Collection and Storage of Umbilical Cord Blood for Transplantation
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LAB04-0249; R01CA061508 (NIH)
Record Dates: First submitted 2012-11-09; First posted 2012-11-20 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Cord Blood Stem Cell Transplantation; Cord Blood Transplantation; Hematopoietic Stem Cell Transplantation
Keywords: Cord blood registry; Umbilical Cord Blood; fetal blood; placenta; Placental Blood Stem Cell Transplantation; hematopoietic progenitor cells; Hematopoietic Stem Cell Transplantation; cord blood unit total nucleated cell; TNC; CD34-positive(+) cell; human leukocyte antigen; HLA; allogeneic transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples from the umbilical cords of newborn babies, a minimum of 40 ml is needed for processing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to collect blood samples from the umbilical cords of newborn babies, as soon as they are delivered, and to place these samples in the MD Anderson Cord Blood Bank. Your sample may be included in the National Cord Blood Inventory (NCBI) which is part of the CW Bill Young Cell Transplantation Program. The NCBI is a federally-supported program to assist in the collection of cord blood. Cord blood will be made available to patients through The National Marrow Donor Program (NMDP). These samples may then be offered to MD Anderson and other institutions for patients who need a bone marrow transplant and do not have a donor. The MD Anderson Cord Blood Bank will have the rights to release cord blood units to these institutions around the world according to established bone marrow transplant donor criteria, for a fee to cover costs.

Cord blood samples that are collected and then do not meet the clinical requirements for patient use may also be used at MD Anderson or other institutions either for research or for quality purposes to improve cord blood banking procedures. If not suitable for patient use or for research purposes, the cord blood unit may be thrown away.

DETAILED DESCRIPTION:
The blood in an unborn baby's umbilical cord contains blood-making cells that could help treat another person with a life-threatening disease. These cord blood cells may provide cells for transplants given to patients with marrow diseases such as leukemia. These cord blood transplants can be done when a patient's cell type (human leukocyte antigen, or HLA, type) matches the cord blood type. 'Cord blood' is normally thrown away with the umbilical cord and placenta after the baby is born.

Collection of the cord blood takes place after your new baby is born and the umbilical cord has been clamped and cut in the normal way. The collection of cord blood takes place from the part of the cord that is still connected to the placenta, not to your new baby. The cord blood may be collected 'in-utero': after your baby is delivered but the placenta is still inside the uterus, or it may be collected 'ex-utero': after the placenta is delivered. The choice of which method of collection is performed will depend on the preference of your obstetrician/midwife. Neither method puts you or your baby at any risk of injury. Once the cord blood is drawn, it becomes the property of the MD Anderson Cord Blood Bank, and you will not retain any residual interests or rights to this sample.

During the delivery of your baby, your obstetrician has your health and that of your newborn baby as his or her main concern. If you agree to take part in this study, your doctor and/or the Cord Blood Bank staff will try to collect the cord blood, but your doctor's main concern will be the well being of you and your baby. Circumstances may arise which prevent the collection of your cord blood.

The cord blood that is collected will be taken to the MD Anderson Cord Blood Bank Laboratory, where it will be tested or sent out for testing to laboratories accredited for doing those tests as described below.

Just like the donation of blood for transfusion, it is important that cord blood does not carry any infections that can be passed on. When volunteers donate blood to a blood bank, they are asked to fill out a confidential questionnaire about their risks for some infections (like acquired immunodeficiency syndrome (AIDS) caused by the human immunodeficiency virus (HIV), hepatitis, and/or malaria). You will be asked questions like these in a questionnaire. You will also be asked some questions about your family medical history, to check for the chance of an inherited disease that could be passed on with the cord blood. This questionnaire will be completed within 48 hours of your baby being born, and will take about 15 minutes to complete. This questionnaire is used for screening purposes, and may result in your cord blood not being suitable for patient use, in which case the cord blood may be used for research purposes, for quality purposes (to improve cord blood banking procedures), or discarded. Your medical chart, and that of your infant, will be reviewed to help determine whether you may have a disease which could be inherited and thus transmitted with the cord blood to a transplant patient who receives it. Additionally, you will be asked about your family ethnic/racial background; this information is used to help match the cord blood to the patients.

A blood sample (about 2 tablespoonfuls) will be drawn from you to test for infectious diseases including HIV, human T cell Iymphotrophic virus (HTLV), Hepatitis B and C, cytomegalovirus (CMV), West Nile Virus (WNV), Trypanosoma cruzi (T cruzi, a parasitic organism that causes Chagas disease) and syphilis. The cord blood unit itself may also be tested for HIV, HTLV, Hepatitis B and C, CMV, WNV, T. cruzi, syphilis, for bacterial and fungal infection, and for the blood type (ABO/Rh). This testing will be performed at accredited testing laboratories. Small samples of your blood and the cord blood (about 2 teaspoonfuls each) will also be frozen and stored separately to screen for diseases in the future.

If you are delivering your baby in Texas, as per Texas state law, a blood sample will be taken from your baby by the hospital staff and will be sent to the Department of State Health Services to be tested for inherited diseases, known as 'Newborn Screening'. You will be asked to sign a release form which will allow the Department of State Health Services to release these Newborn screening results to the MD Anderson Cord Blood Bank. Since such diseases may be passed on through transplant, your donated cord blood unit will not be banked if positive results are received. The Department of State Health Services will notify your physician of positive or unclear Newborn screening results.

In addition, the cord blood unit and sometimes the maternal blood sample will be tested for its HLA type which will be used to identify matches with the transplant patient who needs the cord blood. This testing will be performed at MD Anderson. A small sample of the cord blood unit will be sent to the Stemcyte and City of Hope Laboratories in California for more sophisticated typing to determine whether the cord blood unit might be useful in treating AIDS patients.

Both your blood and your cord blood are tested for infections, because there are rare instances where an infection could be found in the mother's blood and yet it has not been found in the cord blood. It is also possible although uncommon, that an infection could be found in the cord blood but not in the mother's blood. If the volume of your donated cord blood is not large enough for banking, testing may not be performed.

All information you provide, as well as the identity of you and your new baby will be kept as confidential as possible, to the fullest extent allowed by law. While the MD Anderson Cord Blood Bank has to maintain a link between the cord blood unit and information identifying you, multiple levels of security will protect this. When the information and blood samples are collected, they will be given a unique sample number. Nobody except the Principal Investigator and those designated by the Principal Investigator will have access to any of your personal information. If your cord blood is released to another institution for transplant, there will be no way to determine you were the donor as we keep your identity anonymous. If your donated cord blood cells are used in a transplant, the recipient of your cord blood cells will not be able to access any of your personal information.

At the time of donation, you will be asked to provide MD Anderson Cord Blood Bank an address for you and your physician. If any unclear or positive results are found during the testing of your blood or the cord blood (such as HIV, HTLV, Hepatitis B, Hepatitis C, WNV, Chagas and/or syphilis), the MD Anderson Cord Blood Bank will notify your physician using the information you have provided to the Cord Blood Bank. As required by Texas law a confirmed positive or unclear test for HIV/AIDS or syphilis from your blood or the cord blood will be reported to the Texas Department of State Health Services. Additionally, the Houston Department of Health and Human Services will be notified of any positive West Nile Virus results, and they may contact you to conduct a confidential interview to help track community risk to WNV.

The Cord Blood Bank may also contact you directly, using the contact information you provide, in order to obtain updated information about your child's health regarding inherited disorders and/or communicable diseases, or to request additional information or clarification of information contained in the Cord Blood Bank file. If you become aware of any changes in your baby's health which may affect the suitability of the donated cord blood unit for transplantation, it is important that you contact the Cord Blood Bank at 713-563-8000.

The cord blood will be tested and frozen. Cord blood units that meet clinical specifications will be stored in the MD Anderson Cord Blood Bank, listed on the stem cell donor registries and may be released to MD Anderson or other institutions in the US or around the world following established criteria for bone marrow transplant donors, for a fee to cover handling charges. These institutions will use the cord blood for patients needing a bone marrow transplant. Any fresh or stored cord blood units donated to the Cord Blood Bank that do not meet all the clinical specifications (for example, if they are too small or have bacterial contamination), and cannot be used for patients needing a bone marrow transplant, they may be discarded or used for research or in studies to improve the cord blood banking procedures, either at MD Anderson or at other institutions. Before your cord blood can be used for research, the people doing the research must get specific approval from the Institutional Review Board (IRB) of MD Anderson or the IRB of the institution where the research will be performed. The IRB is a committee made up of doctors, researchers, and members of the community. The IRB is responsible for protecting the participants involved in research studies and making sure all research is done in a safe and ethical manner. All research performed at MD Anderson, including research involving your cord blood from this bank, must first be approved by the IRB.

The cord blood units will be used on a first come, first served basis. At the time of donation, you will be given the address and phone number of the MD Anderson Cord Blood Bank. In the unlikely event that you or another immediate family member develop a disease which would require the use of your donated cord blood, it may be released to you on the same basis that it would be provided to other qualifying patients, if it is still under the control of the MD Anderson Cord Blood Bank and has not already been committed to a patient. You should contact the MD Anderson Cord Blood Bank within one month of collection if you wish to have your donated cord blood unit destroyed. If requested, the research staff will destroy your cord blood unit if it has not been used for research, Cord Blood Bank validation studies or quality control. After this one month period has passed, your cord blood unit will be made available for patient use and you will be unable to request that it be destroyed.

This is an investigational study.

Up to 250,000 women will take part in this study. All will be enrolled through MD Anderson.

ELIGIBILITY:
Inclusion Criteria

1. Pregnant women age 18 or older. Cord blood will not be collected from a minor.
2. Able to give verbal informed consent prior to collection of the cord blood.
3. Able to give written informed consent prior to collection of the cord blood.
4. Willing to provide a personal and family medical history (if available) of herself and the biologic father (if available), prior to or following collection of the cord blood.
5. Willing to consent to testing of her blood and the cord blood for infectious diseases, including human immunodeficiency virus (HIV), human T cell lymphotrophic virus (HTLV), hepatitis B and C, cytomegalovirus (CMV), syphilis (RPR), Trypanosoma cruzi (Chagas) and West Nile Virus (WNV). Incomplete tests or positive infectious disease testing results may result in the cord blood unit being deemed unacceptable for clinical use.
6. Willing to consent to testing the cord blood for HLA type, ABO/RhD type, newborn screening and microbial cultures.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neonates delievered by women age 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 250000 (Estimated)
Dates: Start 2005-04 (Actual); Primary Completion 2099-04 (Estimated); Study Completion 2099-04 (Estimated)

PRIMARY OUTCOMES:
Public Cord Blood Banking | 10 years
  Collection and storage of umbilical cord blood units from normal donors for banking and ultimate transplantation into patients.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shpall, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cord Blood Bank Collection Sites, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org